CLINICAL TRIAL: NCT03508635
Title: A Phase I Adaptive Dose, Double-Blind, Placebo-Controlled, SAD and MAD Study to Measure the Safety, Tolerability, Pharmacokinetics and Pharmacological Effects of Orally Administered CORT125134 in Healthy Subjects
Brief Title: CORT125134 Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CORT125134-120; 2014-001951-21 (EudraCT Number)
Record Dates: First submitted 2017-02-21; First posted 2018-04-26 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Glucocorticoid receptor; antagonist
MeSH Terms: interventions — relacorilant; Mifepristone; Prednisone; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SAD Cohorts 1 through 6 (Experimental): Participants will receive single doses of 5 mg up to 400 mg of CORT125134 (capsule) in a dose escalation format. The doses selected will be subject to amendment based on emerging data.
  Interventions: Drug: CORT125134
- SAD Cohorts 1 through 6 Placebo (Placebo Comparator): Participants will receive single doses of Matching Placebo of CORT125134 (capsule).
  Interventions: Drug: Matching Placebo of CORT125134
- Food Effect Cohort 7 (Experimental): Participants will receive a single dose of CORT125134 (capsule) with a standard high fat breakfast. The dose will be chosen such that it has been previously administered in a prior SAD cohort.
  Interventions: Drug: CORT125134
- Pharmacological Effect Cohort 8 (Experimental): Participants will receive a single dose of 25 mg of prednisone on Day -19; a single dose of 25 mg prednisone and 600 mg of mifepristone on Day -12; and a single dose of 25 mg prednisone and a single dose of CORT125134 on Day 1. The dose of CORT125134 will be chosen such that it has been previously administered in a prior SAD cohort.
  Interventions: Drug: CORT125134; Drug: Mifepristone; Drug: Prednisone
- Proof of Concept (POC) Cohort 9 (Experimental): Participants will receive a single dose of 25 mg of prednisone on Day -19; a single dose of 25 mg of prednisone and 600 mg of mifepristone on Day -12; and a single dose of 25 mg prednisone and a single dose of CORT125134 on Day 1. An oral glucose tolerance test will be administered on each study day. The dose of CORT125134 will be chosen such that it has been previously administered in a prior SAD cohort.
  Interventions: Drug: CORT125134; Drug: Mifepristone; Drug: Prednisone; Drug: Glucose
- MAD Cohorts 10 and 11 (Experimental): Participants will receive the selected dose of CORT125134 (capsule) following receipt of data from Cohorts 1-9 up to a maximum frequency of twice a day for a total of 14 days.
  Interventions: Drug: CORT125134
- MAD Cohorts 10 and 11 Placebo (Placebo Comparator): Participants will receive Matching Placebo of CORT125134 (capsule) up to a maximum frequency of twice a day for a total of 14 days.
  Interventions: Drug: Matching Placebo of CORT125134
- MAD of PoPE Cohorts 12 and 13 (Experimental): Proof of Pharmacological Effect (PoPE+POC). Participants will receive 25 mg of prednisone (both cohorts) and an oral glucose tolerance test (Cohort 13 only) on Day -5. Participants will then receive the selected dose of CORT125134 (capsule) for a total of 13 days. Participants may either receive a higher dose level than previously administered or a repeat of a dose level given in 1 of the previous 2 MAD Cohorts. Participants will then receive 25 mg of prednisone (both cohorts) and an oral glucose tolerance test (Cohort 13 only) on Day 14.
  Interventions: Drug: CORT125134; Drug: Prednisone; Drug: Glucose
- MAD of PoPE Cohort 12 and 13 Placebo (Placebo Comparator): Participants will receive 25 mg of prednisone (both cohorts) and an oral glucose tolerance test (Cohort 13 only) on Day -5. Participants will then receive the Matching Placebo of CORT125134 (capsule) for a total of 13 days. Participants will then receive 25 mg of prednisone (both cohorts) and an oral glucose tolerance test (Cohort 13 only) on Day 14.
  Interventions: Drug: Matching Placebo of CORT125134; Drug: Prednisone; Drug: Glucose

INTERVENTIONS:
Drug: CORT125134 — Oral capsules
  Arms: Food Effect Cohort 7; MAD Cohorts 10 and 11; MAD of PoPE Cohorts 12 and 13; Pharmacological Effect Cohort 8; Proof of Concept (POC) Cohort 9; SAD Cohorts 1 through 6
Drug: Matching Placebo of CORT125134 — Placebo
  Arms: MAD Cohorts 10 and 11 Placebo; MAD of PoPE Cohort 12 and 13 Placebo; SAD Cohorts 1 through 6 Placebo
Drug: Mifepristone — Active comparator
  Arms: Pharmacological Effect Cohort 8; Proof of Concept (POC) Cohort 9
Drug: Prednisone — Challenge agent
  Arms: MAD of PoPE Cohort 12 and 13 Placebo; MAD of PoPE Cohorts 12 and 13; Pharmacological Effect Cohort 8; Proof of Concept (POC) Cohort 9
Drug: Glucose
  Arms: MAD of PoPE Cohort 12 and 13 Placebo; MAD of PoPE Cohorts 12 and 13; Proof of Concept (POC) Cohort 9

SUMMARY:
The purpose of this study is to evaluate the dose-related safety, tolerability, pharmacokinetics (PK) and pharmacological effects (PD) of CORT125134 and its active metabolite CORT125201 after single and multiple ascending oral doses of CORT125134 in healthy participants.

DETAILED DESCRIPTION:
This is a 3-part, single-center study of single and multiple ascending doses of CORT125134 in healthy participants.

Part I is a single dose study. Initially, participants will be enrolled sequentially into 1 of up to 6 cohorts, each containing 10 participants, in a double-blind, randomized, placebo-controlled assessment of single-ascending doses (SAD) of CORT125134. Within each cohort, 8 participants will be randomly assigned to receive a single dose of CORT125134, and 2 participants will be randomly assigned to receive a single dose of matching placebo. Thereafter, Cohort 7 will be a food-effect cohort, in which all 8 participants will receive a single dose of CORT125134 after a high-fat breakfast (open label). Cohorts 8 and 9 will be pharmacological effect cohorts, in each of which 10 participants will receive a challenge agent (prednisone, 25 mg) alone on Day -19; with an active comparator (mifepristone, 600 mg) on Day -12, and with CORT125134 on Day 1 in an open-label single sequence crossover design. Pharmacological effects will be explored by measuring effects on peripheral blood eosinophil, lymphocyte and neutrophil counts, serum osteocalcin, assay of messenger ribonucleic acid (mRNA) expression of FK506 Binding Protein 5 (FKBP5) and Glucocorticoid-induced Leucine Zipper (GILZ) in whole blood (proof of pharmacological effect Cohort 8) and by measuring effects on oral glucose tolerance (proof of concept Cohort 9).

Part 2 and 3 will be double-blind, randomized, placebo-controlled assessments of multiple oral ascending doses (MAD) of CORT125134. Participants will be enrolled sequentially into 1 of up to 4 cohorts (Cohorts 10-13), each containing 12 participants. Within each cohort, 9 participants will be randomly assigned to receive CORT125134 and 3 participants to receive matching placebo daily for 14 days (Days 1-14). The effects of CORT125134 on response to prednisone challenge will be additionally explored in Cohorts 12 and 13 in a single sequence crossover, with prednisone being given alone on Day -5 and in combination with CORT125134 or placebo on Day 14.

Throughout the study, routine safety tests and assessments of PK (CORT125134 and CORT125201) will be performed, and changes in serum cortisol and plasma adrenocorticotrophic hormone (ACTH) measured.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Weight <= 102 kilogram (kg); body mass index (BMI) 18-30 kg/meter squared
* Morning serum cortisol in reference range
* Willing and able to communicate, participate in the whole study and to abide by study restrictions including use of contraception

Exclusion Criteria:

* Participation in any clinical research study, received treatment with any investigational drug or device, or donated blood within the previous 3 months
* Has a history of alcoholism, substance abuse, or drug abuse within 1 year; positive screen for alcohol or drugs of abuse
* Current smokers, smoked and/or used tobacco and/or nicotine-containing products within 6 months, or positive screen for carbon monoxide
* Females of childbearing potential, pregnant or breastfeeding, and/or with a positive pregnancy test
* Has a condition that could be aggravated by glucocorticoid blockade or activation
* Has clinically relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead electrocardiogram (ECG)
* Has history of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, chronic respiratory, gastrointestinal or neurological disease
* Has used systemic glucocorticoids within 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) (Safety and Tolerability) of CORT125134 | Single dose Cohorts 1-9 Day 1 to Day 15; MAD Cohorts 10-13 Day 1 to Day 28/Day 24 (Cohort 13)

SECONDARY OUTCOMES:
QT internal corrected for heart rate using Fridericia's formula (QTcF) exposure-response analysis | SAD Cohorts 1-6: Pre dose through 24 hours post dose; MAD Cohorts: Pre first dose through 24 hours post final dose of Investigational Medicinal Product (IMP)
CORT125134 Pharmacokinetic (PK) of total lag time (Tlag) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Day 28/24 (Cohort 13)
CORT125134 PK of peak plasma concentration (Cmax) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Day 28/24 (Cohort 13)
CORT125134 PK of time to reach maximum observed concentration (Tmax) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts 10-12 Day 1 to Day 28/24 (Cohort 13)
CORT125134 PK of area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUClast) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Day 28/24 (Cohort 13)
CORT125201 PK of peak plasma concentration (Cmax) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Day 28/24 (Cohort 13)
CORT125201 PK time Lag (Tlag) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Day 28/24 (Cohort 13)
CORT125201 PK of time to reach maximum observed concentration (Tmax) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Day 28/24 (Cohort 13)
CORT125201 PK of area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUClast) | Single dose Cohorts Day 1 to Day 15; MAD Cohorts Day 1 to Say 28/24 (Cohort 13)
Eosinophil count | Single dose Cohort 8 Days -19 to Day 2; MAD Cohorts 12 and 13 Days -5 to Day 15
Lymphocyte count | Single dose Cohort 8 Days -19 to Day 2; MAD Cohorts 12 and 13 Days -5 to Day 15
Neutrophil count | Single dose Cohort 8 Days -19 to Day 2; MAD Cohorts 12 and 13 Days -5 to Day 15
Osteocalcin | Single dose Cohort 8 Days -19 to Day 2; MAD Cohorts 12 and 13 Days -5 to Day 15
FKBP5 expression | Single dose Cohort 8 Days -19 to Day 2; MAD Cohorts 12 and 13 Days -5 to Day 15
Glucocorticoid-induced leucine zipper (GILZ) expression | Single dose Cohort 8 Days -19 to Day 2; MAD Cohorts 12 and 13 Days -5 to Day 15
Glucose tolerance | Single dose Cohort 9 Days -19 to Day 2; MAD Cohort 13 Days -5 to Day 15
Serum cortisol | SAD Cohorts 1-6: Pre dose to Day 15; MAD Cohorts 10-11: Pre dose to Day 28
Plasma adrenocorticotrophic hormone (ACTH) | SAD Cohorts 1-6: Pre dose to Day 15; MAD Cohorts 10-11: Pre dose to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hunt H, Donaldson K, Strem M, Zann V, Leung P, Sweet S, Connor A, Combs D, Belanoff J. Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacological Effect of Orally Administered CORT125134: An Adaptive, Double-Blind, Randomized, Placebo-Controlled Phase 1 Clinical Study. Clin Pharmacol Drug Dev. 2018 May;7(4):408-421. doi: 10.1002/cpdd.389. Epub 2017 Oct 2. PMID 28967708